CLINICAL TRIAL: NCT04532281
Title: Clinical Trial for the Safety and Efficacy of Murine CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia and B-cell Non-Hodgkin's Lymphoma
Brief Title: A Study of Murine CD19 CAR-T Therapy for Patients With Relapsed or Refractory CD19+ B-cell Hematological Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mCD19-002
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin Lymphoma of Soft Tissue
Keywords: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; CAR T-cell therapy; CD19
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Murine CD19 CAR T-cells (Experimental)
  Interventions: Drug: Murine CD19 CAR-T cells

INTERVENTIONS:
Drug: Murine CD19 CAR-T cells — Each subject receive murine CD19 CAR T-cells by intravenous infusion
  Other Names: Murine CD19 CAR-T cells injection

SUMMARY:
A Study of Murine CD19 CAR-T Cells Therapy for Patients With Relapsed or Refractory CD19+ B-cell Hematological Malignancies.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD19+ B-cell hematological malignancies, including acute lymphoblastic leukemia and B-cell non-Hodgkin's lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. Two groups of patients will be enrolled, 36 in each group. Primary objective is to explore the safety, main consideration is dose- related safety.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria only for B-ALL:

  1. Histologically confirmed diagnosis of CD19+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1)；
  2. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

     1. CR not achieved after standardized chemotherapy;
     2. CR achieved following the first induction, but CR duration is less than 12 months;
     3. Ineffectively after first or multiple remedial treatments;
     4. 2 or more relapses;
  3. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is > 5% (by morphology), and/or > 1% (by flow cytometry);
  4. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;
* Inclusion criteria only for B-NHL:

  1. Histologically confirmed diagnosis of DLBCL (NOS), FL, DLBCL transformed from CLL/SLL, PMBCL, and HGBCL per the WHO Classification Criteria for Lymphoma (2016);
  2. Relapsed or refractory B-NHL (meeting one of the following conditions):

     1. No response or relapse after second-line or above chemotherapy regimens;
     2. Primary drug resistance;
     3. Relapse after auto-HSCT;
  3. At least one assessable tumor lesion per Lugano 2014 criteria;
* Common inclusion criteria for B-ALL and B-NHL:

  1. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
  2. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
  3. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
  4. Estimated survival time ≥ 3 months;
  5. ECOG performance status 0 to 2;
  6. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance, epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tractinfectionand bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
7. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after murine CD19 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after murine CD19 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia(B-ALL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
B-ALL, Overall survival (OS) | Up to 2 years after murine CD19 CAR-T cells infusion
  From the first infusion of murine CD19 CAR-T cells to death or the last visit
B-ALL, Event-free survival (EFS) | Up to 2 years after murine CD19 CAR-T cells infusion
  From the first infusion of murine CD19 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | At Week 4, 12, and Month 6, 12, 18, 24
  Assessment of ORR (ORR = CR + PR) per Lugano 2014 criteria
B-NHL, disease control rate (DCR) | At Week 12 and Month 6, 12, 18, 24
  Assessment of DCR (DCR=CR+PR+SD) per Lugano 2014 criteria
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No